CLINICAL TRIAL: NCT00013247
Title: Facilitating Shared Decisionmaking About Prostate Cancer Screening
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 99-277
Record Dates: First submitted 2001-03-14; First posted 2001-03-16 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2007-02

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Other)
  Interventions: Behavioral: Prostate Cancer Screening Education

INTERVENTIONS:
Behavioral: Prostate Cancer Screening Education

SUMMARY:
Due to the disputed efficacy of prostate cancer (CaP) screening and treatment, most authorities recommend that providers inform and involve patients in CaP screening decisions.

DETAILED DESCRIPTION:
Background:

Due to the disputed efficacy of prostate cancer (CaP) screening and treatment, most authorities recommend that providers inform and involve patients in CaP screening decisions.

Objectives:

This study evaluated two interventions designed to facilitate this process.

Methods:

1152 male veterans age 50+ with no CaP and primary care appointments at four VA medical facilities in VISN 23 were randomly assigned to one of three groups: mailed pamphlet intervention, mailed video intervention, or usual care (control). Intervention materials were mailed two weeks prior to a target primary care appointment and patient telephone surveys were conducted one week (T1) and one year (T2) after the target appointment. Outcomes included: a 10- item validated knowledge index; responses to questions on CaP natural history, treatment efficacy, PSA accuracy, and expert disagreement about the PSA; whether screening was discussed with provider; scores on decision information seeking, participation and satisfaction scales; screening and treatment preferences; and PSA testing rates.

Status:

Complete

ELIGIBILITY:
Inclusion Criteria:

Patients must be male veterans, age 50 and older, with a scheduled primary care appointment at one of 5 VISN 13 medical facilities. Patients diagnosed with prostate cancer will be excluded.

Exclusion Criteria:

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1152 (Estimated)
Dates: Study Completion 2002-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa R. Partin, PhD, Principal Investigator — Minneapolis VA Health Care System, Minneapolis, MN
Locations (1):
- Minneapolis VA Health Care System, Minneapolis, MN, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Partin MR, Nelson D, Flood AB, Friedemann-Sanchez G, Wilt TJ. Who uses decision aids? Subgroup analyses from a randomized controlled effectiveness trial of two prostate cancer screening decision support interventions. Health Expect. 2006 Sep;9(3):285-95. doi: 10.1111/j.1369-7625.2006.00400.x. PMID 16911143
- [Result] Radosevich DM, Partin MR, Nugent S, Nelson D, Flood AB, Holtzman J, Dillon N, Haas M, Wilt TJ. Measuring patient knowledge of the risks and benefits of prostate cancer screening. Patient Educ Couns. 2004 Aug;54(2):143-52. doi: 10.1016/S0738-3991(03)00207-6. PMID 15288907
- [Result] Wilt TJ, Partin MR. Reducing PSAnxiety: The importance of noninvasive chronic disease management in prostate cancer detection and treatment. Am J Med. 2004 Nov 15;117(10):796-8. doi: 10.1016/j.amjmed.2004.10.002. No abstract available. PMID 15541329
- [Result] Wilt TJ, Partin MR. Prostate cancer intervention. Involving the patient in early detection and treatment. Postgrad Med. 2003 Oct;114(4):43-9; quiz 50. doi: 10.3810/pgm.2003.10.1506. PMID 14587206
- [Result] Partin MR, Nelson D, Radosevich D, Nugent S, Flood AB, Dillon N, Holtzman J, Haas M, Wilt TJ. Randomized trial examining the effect of two prostate cancer screening educational interventions on patient knowledge, preferences, and behaviors. J Gen Intern Med. 2004 Aug;19(8):835-42. doi: 10.1111/j.1525-1497.2004.30047.x. PMID 15242468
- [Result] Taylor BC, Wilt TJ, Clothier B, Grill JP, Partin MR. Assessing health status in older men with lower urinary tract symptoms. Federal practitioner : for the health care professionals of the VA, DoD, and PHS. 2006 Jul 1; 23(7):29-40.